CLINICAL TRIAL: NCT06940557
Title: Evaluating The Efficacy And Tolerability Of The Oral Combination Of Alpha Lipoic Acid And Vitamin B Complex Preparation In Carpal Tunnel Syndrome : a Single-center, Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Efficacy And Tolerability Of Alpha Lipoic Acid And Vitamin B Preparation In Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: BREGO Life Sciences Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Anna Misyail Abdul Rashid, Dr,, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JKEUPM-2022-984
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Vitamin B; Alpha Lipoic Acid; CTS; NCS; BCTQ; SF-36; VAS
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treament (Active Comparator): alpha lipoic acid; 300mg, methylcobalamin; 500mcg, vitamin B1; 39mg and vitamin B6; 8mg 2 tablets once daily
  Interventions: Drug: Bionerv
- Placebo (Placebo Comparator): maltodextrin, microcrystalline cellulose, tricalcium phosphate, silicon gioxide, magnesium stearate 2 tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bionerv — alpha lipoic acid; 300mg, methylcobalamin; 500mcg, vitamin B1; 39mg and vitamin B6; 8mg, 2 tablets once daily
  Other Names: Group A
  Arms: Treament
Drug: Placebo — maltodextrin, microcrystalline cellulose, tricalcium phosphate, silicon gioxide, magnesium stearate 2 tablets once daily
  Other Names: Group B
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the effectiveness and safety of an oral combination of alpha lipoic acid (ALA) and vitamin B complex in treating mild to moderate carpal tunnel syndrome (CTS) in adults. The main questions it aims to answer are:

* Does the combination of ALA and vitamin B improve nerve function (based on electrodiagnostic studies) in patients with CTS?
* Does this treatment reduce CTS-related symptoms and improve quality of life?
* What side effects, if any, do participants experience while taking the treatment?

Researchers will compare the combination of ALA and vitamin B to a placebo (a look-alike substance that contains no active drug) to evaluate its effectiveness.

Participants will:

* Take the ALA and vitamin B combination or a placebo once daily for 6 months.
* Attend clinic visits at the start of the study, after 3 months, and after 6 months for physical examinations, nerve conduction studies, and to complete questionnaires about their symptoms and quality of life.
* Receive follow-up phone calls and reminder messages to ensure medication compliance and attendance at scheduled visits.

DETAILED DESCRIPTION:
The patients were randomized to receive oral combination of alpha lipoic acid and vitamin B (alpha lipoic acid; 300mg, methylcobalamin; 500mcg, vitamin B1; 39mg and vitamin B6; 8mg), 2 tablets once daily or placebo drug (maltodextrin, microcrystalline cellulose, tricalcium phosphate, silicon gioxide, magnesium stearate) 2 tablets once daily. Randomization sequence was done by using an online random number generator program using a mixed block randomization technique at a ratio of 1:1. In cases of serious adverse event, unblinding process was incorporated where the identity of the drug was revealed to manage the subject's condition. This was done by intruding the emergency code key by the researcher. All patients provided a written consent for the study.

During visit 1, a thorough history and physical examination were done, and demographic data was collected. Afterward, the patients were required to answer three sets of self-administered questionnaires: Boston Carpal Tunnel Questionnaire (BCTQ), Visual analogue score (VAS) and SF-36. The BCTQ is a specific questionnaire for assessing CTS that consists of two distinct scales, the Symptom Specific Scale (SSS) which has 11 items and the Functional Status Scale (FSS) containing 8 items. Each scale generates a final score ranging from 1 to 5, with a higher score indicating greater disability and poor symptoms control. BCTQ is a reliable questionnaire to assess CTS owing to its high cross-cultural adaptation and multilingual validity and reliability. The VAS is a visual scale with 0 scored as "no pain" and 10 as "worst pain imaginable" and serves as an excellent tool for pain score with excellent validity and reproducibility. The SF-36 is a quality-of-life questionnaire that comprises of 36 questions covering eight domains of health which are; Physical Functioning (PF), Role Limitations due to Physical Health, Role Limitations (RL) due to Emotional Problems (RE), energy/fatigue, emotional well-being, social functioning, pain, and general health (GH) where a higher score indicates a better outcome . After the administration of these questionnaires, they will be subjected for a nerve conduction study (NCS) to determine the severity of CTS. The NCS were performed by the same trained personnel to ensure consistency and accuracy.

The patients were reassessed at Visit 2 (3 months post-treatment) and Visit 3 (6 months post-treatment). During each visit, they underwent physical examination, NCS, and were required to complete the three sets of questionnaires (BCTQ, VAS, and SF-36). They were also required to fill in the form regarding the side effects of the treatments. The investigators made a phone call and sent reminder message at the 6th and 18th week to ensure compliance, medication adequacy and follow up review. During the study, patients were allowed to undergo the standard of care treatment at our center such as physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* all patients with numbness and tingling sensation at the first finger until the radial site of the 4th finger
* and/or fulfil the electrodiagnostic criteria of mild to moderate CTS, based on the Padua Scale as defined below:

  * Mild: abnormal digit/wrist Sensory Nerve Conduction Velocity (CV) and normal Distal Motor Latency (DML)
  * Moderate: abnormal digit/wrist Sensory Nerve Conduction Velocity (SNCV) and abnormal Distal Motor Latency (DML).

Exclusion Criteria:

* pregnant or breastfeeding women
* patients with symptoms of CTS but have normal NCS
* patients taking traditional or complementary medication for CTS
* patients with electrodiagnostic criteria of severe or extreme CTS as defined in the Padua scale:

  * Severe: Absence of sensory response (SNAP) and abnormal Distal Motor Latency (DML).
  * Extreme: Absence of motor (CMAP) and sensory responses (SNAP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement on Nerve Conduction Study | Enrolment (Visit 0) to Visit 1 (3 months) and to Visit 2 (6 months)
  Electrodiagnostic improvement of the median nerve on Nerve Conduction Study (NCS)

SECONDARY OUTCOMES:
Improvements in symptoms using the Boston Carpal Tunnel Questionnaire (BCTQ) | Enrolment (Visit 0) to Visit 1 (3 months) and to Visit 2 (6 months)
  The BCTQ is a specific self administered questionnaire for assessing CTS that consists of two distinct scales, the Symptom Specific Scale (SSS) which has 11 items and the Functional Status Scale (FSS) containing 8 items. Each scale generates a final score ranging from 1 to 5, with a higher score indicating greater disability and poor symptoms control. BCTQ is a reliable questionnaire to assess CTS owing to its high cross-cultural adaptation and multilingual validity and reliability
Improvements in symptoms using the visual analog score (VAS) | Enrolment (Visit 0) to Visit 1 (3 months) and to Visit 2 (6 months)
  The VAS is a visual scale with 0 scored as "no pain" and 10 as "worst pain imaginable" and serves as an excellent tool for pain scoring with excellent validity and reproducibility
Improvements in quality of life using the SF-36 questionnaire | Enrolment (Visit 0) to Visit 1 (3 months) and to Visit 2 (6 months)
  The SF-36 is a quality-of-life is a self administered questionnaire that comprises 36 questions covering eight domains of health: physical functioning (PF), role limitations due to physical health, role limitations (RL) due to emotional problems (RE), energy/fatigue, emotional well-being, social functioning, pain, and general health (GH), where a higher score indicates a better outcome.

OTHER OUTCOMES:
Side effects of the treatment and tolerability | Enrolment (Visit 0) to Visit 1 (3 months) and to Visit 2 (6 months)
  The tolerability in this study is based on patient reporting side-effects that developed after taking the medications using a self-administered reporting form. There are no blood or radiological investigation involved to confirm its association with the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: ANNA MISYAIL ABDUL RASHID, NEUROLOGIST, Principal Investigator — UPM
Locations (1):
- Hospital Sultan Abdul Aziz Shah, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared to ensure patient confidentiality, as participants did not provide explicit consent for data sharing. Additionally, ethical guidelines, regulatory constraints, and concerns about potential data misuse further limit the feasibility of sharing IPD.

REFERENCES:
- [Background] Padua L, LoMonaco M, Gregori B, Valente EM, Padua R, Tonali P. Neurophysiological classification and sensitivity in 500 carpal tunnel syndrome hands. Acta Neurol Scand. 1997 Oct;96(4):211-7. doi: 10.1111/j.1600-0404.1997.tb00271.x. PMID 9325471
- [Background] Di Geronimo G, Caccese AF, Caruso L, Soldati A, Passaretti U. Treatment of carpal tunnel syndrome with alpha-lipoic acid. Eur Rev Med Pharmacol Sci. 2009 Mar-Apr;13(2):133-9. PMID 19499849
- [Background] Passiatore M, Perna A, De-Vitis R, Taccardo G. The Use of Alfa-Lipoic Acid-R (ALA-R) in Patients with Mild-Moderate Carpal Tunnel Syndrome: A Randomised Controlled Open Label Prospective Study. Malays Orthop J. 2020 Mar;14(1):1-6. doi: 10.5704/MOJ.2003.001. PMID 32296475

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06940557/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06940557/ICF_001.pdf